CLINICAL TRIAL: NCT04090502
Title: Effectiveness of Hamstring Muscle Dry Needling in Patients With Chronic Mechanical Low Back Pain of Non-specific Origin
Brief Title: Treatment of Hamstring Muscle in Patients With Low-back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Clinical professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEIM/HU2019/18
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Low Back Pain
Keywords: pain; Back; Hamstrings
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grupo A. Dry needling in Trigger point (Experimental): Participants will be treated in the most hyperalgesic foci within the hamstring musculature.
  Interventions: Other: Dry needling in hamstring muscle trigger points
- Grupo B. Dry needling in non-hyperalgesic areas (Placebo Comparator): Participants will be treated in non-hyperalgesic areas within the hamstring muscles.
  Interventions: Other: Dry needling in hamstring muscle not trigger points

INTERVENTIONS:
Other: Dry needling in hamstring muscle trigger points — Participants with nonspecific mechanical low back pain will be assessed for the hamstring muscle. Subsequently, the most sensitive areas associated with the shortening of the muscle will be located and the technique will be applied to this area.
  Other Names: intramuscular stimulation of muscle
  Arms: Grupo A. Dry needling in Trigger point
Other: Dry needling in hamstring muscle not trigger points — Participants with nonspecific mechanical low back pain will be assessed for the hamstring muscle. Subsequently, the most sensitive areas associated with the shortening of the muscle will be located and the technique will be applied out of this area.
  Arms: Grupo B. Dry needling in non-hyperalgesic areas

SUMMARY:
This study evaluates the treatment of hamstrings in the management of patients with mechanical low back pain of non-specific origin. Half of the participants will received the application of a dry needle technique in the most hyperalgesic areas of the muscle, while the other half will received the same technique in areas not hyperalgesic.

DETAILED DESCRIPTION:
Shortening of the hamstrings could be related to low back pain.Therefore, the treatment of these muscles may improve pain.

The dry needling technique seems to improve the extensibility of the muscles. This technique seems to be more effective when is applied in the most hyperalgesic areas related to the participant's pain.

In order to demonstrate this hypothesis, the investigators will check if the dry needling technique produces the same effects when is applied in other areas of those same muscles

ELIGIBILITY:
Inclusion Criteria:

* Nonspecific chronic low back pain lasting ≥ 3 months.
* Age between 18 and 65 years.
* History of non-specific lumbar pain not irradiated to lower extremities of at least 1 year of evolution.
* Those subjects who have not received a physiotherapy session in the last 6 months.

Exclusion Criteria:

* Specific low back pain (infection, tumor, inflammation, canal stenosis, spondylolisthesis, hernia or disc prolapse, structural deformity, rheumatic disease, radicular pain, cauda equina, previous history of spinal surgery).

  * Fibromyalgia.
  * Treatment with corticosteroids or oral medications in the last 6 months.
  * History of spinal surgery.
  * Contraindications typical of deep dry puncture (needle phobia, coagulation or psychological disorders, varicose regions, cysts, wounds, metal or latex allergy, lymphedema, hypothyroidism, diabetes).
  * Those subjects with a value of 0º in the Active Knee Extension (EAR) test.
  * Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Low back pain | Change from Baseline Pressure Pain Threshold at 3 months
  The investigators use a Visual Analog Scale (VAS) to determine the intensity of the patient with blowback pain.The VAS is a 100-mm line, oriented horizontally, with one end representing "no pain" and the other end representing "worst pain." Subjects will be asked to rate their current pain with a mark on the scale.

SECONDARY OUTCOMES:
Disability with Oswestry Disability Index | Change from Baseline disability at 3 months
  The Oswestry Disability Index (ODI) is a questionnaire used by clinicians and researchers to quantify disability for low back pain.The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel.Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible
The extensibility of the hamstring muscle | Change from Baseline disability at 3 months
  The extensibility of the hamstring muscle will be measured by the popliteal or active knee extension (AKE) test, with the patient supine on the stretcher, with the contralateral limb in extension, will placed with the hip at 90 degrees of flexion.
  While maintaining this position, the clinician tries to extend the knee. Limitation of knee extension is measured with a goniometer in degrees.
Pressure Pain Threshold | Change from Baseline Pressure Pain Threshold at 3 months
  The PPT serves to determine the sensitivity of hiperalgesic focus. The investigators will done it with one algometer. A lower threshold is a worse result. A higher threshold is a better result.

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Gallego-Izquierdo, PhD, Study Chair — Alcala University
Locations (2):
- Spain (2):
  - Centro Investigación Fisioterapia y Dolor, Alcalá de Henares, Madrid
  - Instituto Fisioterapia y Dolor, Alcalá de Henares, Madrid